CLINICAL TRIAL: NCT07290075
Title: The Relationship Between Olfactory and Gustatory Senses, Hedonic Hunger, and Diet Quality After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Hanife Köksal (Other)
Collaborators: Uskudar University (Other)
Responsible Party: Sponsor-Investigator, Hanife Köksal, Registered dietitians, Istanbul University
Organization: Istanbul University (Other)
Other Study IDs: USK-NUTR-HK01
Record Dates: First submitted 2025-08-12; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Taste Disorders; Smell Disorder
Keywords: Hedonic Hunger; bariatric surgery outcomes; Mediterranean Diet; Nutrient Adequacy; Power of Food Scale (PFS); Taste and Smell Questionnaire; MEDAS
MeSH Terms: conditions — Obesity; Taste Disorders; Olfaction Disorders | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sleeve Gastrectomy (SG): Participants who underwent sleeve gastrectomy at least 3 months prior to enrollment.
  Interventions: Other: Sleeve Gastrectomy (SG) and Roux-en-Y Gastric Bypass (RYGB)
- Roux-en-Y Gastric Bypass (RYGB): Participants who underwent Roux-en-Y gastric bypass at least 3 months prior to enrollment.
  Interventions: Other: Sleeve Gastrectomy (SG) and Roux-en-Y Gastric Bypass (RYGB)

INTERVENTIONS:
Other: Sleeve Gastrectomy (SG) and Roux-en-Y Gastric Bypass (RYGB) — Participants who have undergone sleeve gastrectomy ≥3 months prior to study enrollment; and Participants who have undergone Roux-en-Y gastric bypass ≥3 months prior to study enrollment.

SUMMARY:
This cross-sectional observational study investigates the association between changes in olfactory and gustatory senses and hedonic hunger among individuals who have undergone bariatric surgery. The study also examines the effects of these sensory changes on diet quality and anthropometric measurements. Participants completed a structured questionnaire including sociodemographic and health information, dietary habits, a modified 33-item taste and smell assessment, the Power of Food Scale (PFS), the Mediterranean Diet Adherence Screener (MEDAS), the International Physical Activity Questionnaire (IPAQ), and anthropometric measurements.

DETAILED DESCRIPTION:
Obesity is a chronic, multifactorial disease that negatively impacts health and quality of life. Bariatric surgery is an effective treatment option for severe obesity, leading to significant and sustained weight loss as well as improvement in obesity-related comorbidities.

Postoperative changes in taste and smell perception are frequently reported by bariatric patients and may influence food preferences, hedonic hunger, and overall diet quality. These sensory alterations can result from anatomical and hormonal changes after surgery, including altered gut hormone secretion (e.g., PYY, GLP-1, ghrelin) and bile acid metabolism, which affect appetite regulation and reward pathways.

This cross-sectional observational study evaluated adults aged 18-65 years who had undergone sleeve gastrectomy (SG) or Roux-en-Y gastric bypass (RYGB) at least three months prior to enrollment. Data collection included sociodemographic and health information, dietary habits, a modified 33-item taste and smell questionnaire, the Power of Food Scale (PFS) to assess hedonic hunger, the Mediterranean Diet Adherence Screener (MEDAS), the International Physical Activity Questionnaire (IPAQ), and anthropometric measurements. Nutrient intakes were analyzed according to the Türkiye Nutrition Guide (TÜBER-2022) reference values.

The primary objective was to determine the relationship between postoperative taste/smell changes and hedonic hunger. Secondary objectives included assessing the association between sensory perception and Mediterranean diet adherence, anthropometric parameters, and nutrient adequacy by surgery type. Findings from this study may guide the development of personalized nutritional follow-up protocols to improve long-term outcomes in bariatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years
* History of bariatric surgery (Sleeve Gastrectomy or Roux-en-Y Gastric Bypass)
* At least 3 months post-surgery at the time of study enrollment
* Able and willing to provide informed consent

Exclusion Criteria:

* Pregnancy
* History of neurological disorders affecting taste or smell
* Active upper respiratory infection at the time of assessment
* Severe psychiatric disorders that may impair participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-65 years who have undergone bariatric surgery (Sleeve Gastrectomy or Roux-en-Y Gastric Bypass) at least 3 months prior to enrollment, recruited from patients followed in clinical nutrition and bariatric surgery outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Power of Food Scale (PFS) Score | Baseline (Day 1, at study enrollment)
  Hedonic hunger assessed using the Power of Food Scale (range: 1-5; higher scores indicate greater hedonic hunger).
Modified 33-item Taste and Smell Questionnaire Score | Baseline (≥3 months after bariatric surgery, at study enrollment)
  Changes in taste and smell perception assessed using a modified 33-item questionnaire (range: 0-33; higher scores indicate more pronounced sensory changes).

SECONDARY OUTCOMES:
Mediterranean Diet Adherence Screener (MEDAS) Score | Baseline (≥3 months after bariatric surgery, at study enrollment)
  Adherence to the Mediterranean diet assessed using the 14-item MEDAS questionnaire (range: 0-14; higher scores indicate greater adherence).
Body Mass Index (BMI) | Baseline (Day 1, at study enrollment)
  BMI calculated as weight (kg) / height (m²).
Waist-to-Hip Ratio (WHR) | Baseline (Day 1, at study enrollment)
  WHR calculated as waist circumference (cm) / hip circumference (cm).
Energy Intake Adequacy (% of TÜBER-2022 reference) | Baseline (Day 1, at study enrollment)
  Daily energy intake adequacy compared to TÜBER-2022 reference values.
Protein Intake Adequacy (% of TÜBER-2022 reference) | Baseline (Day 1, at study enrollment)
  Daily protein intake adequacy compared to TÜBER-2022 reference values.
Micronutrient Intake Adequacy (e.g., iron, folate, vitamin E; % of TÜBER-2022 reference) | Baseline (Day 1, at study enrollment)
  Micronutrient intake adequacy compared to TÜBER-2022 reference values.
Nutrient Adequacy Score (based on TÜBER-2022 reference values) | Baseline (Day 1, at study enrollment)
  Composite score reflecting the percentage adequacy of daily energy, macronutrient, and micronutrient intakes compared to TÜBER-2022 reference values. Higher scores indicate greater adequacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Faculty of Medicine, Department of Endocrinology and Metabolism, Istanbul, Capa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No - Individual participant data (IPD) will not be shared due to privacy concerns and lack of prior consent for public data sharing from study participants. Only aggregated results will be available in publications.